CLINICAL TRIAL: NCT06763185
Title: Comparative Effects of Conventional Cow's Milk Versus Milk Free of A1-type Beta-casein on Gastrointestinal Physiology and Symptoms of Digestive Discomfort in Participants Intolerant to Conventional Cow's Milk: a Randomised Controlled Trial
Brief Title: A1 Beta-casein-free Milk in Milk-intolerant Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: a2 Milk Company Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Supportive Care
Other Study IDs: 1016-065 Milk
Record Dates: First submitted 2024-12-11; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Digestive Discomfort
Keywords: milk free of A1-type beta-casein; conventional cow's milk; gastrointestinal symptoms

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sequence 1 (Other): Sequence 1: a 2-week washout period, 2 weeks of conventional cow's milk consumption, crossover, a second 2-week washout period, and a second 2-week period of A1PF milk consumption.
  Interventions: Other: Dietary Supplement: conventional cow's milk consumption, and then A1PF milk consumption
- Sequence 2 (Other): Sequence 2: a 2-week washout period, 2 weeks of A1PF milk consumption, crossover, a second 2-week washout period, and a second 2-week period of conventional cow's milk consumption.
  Interventions: Other: Dietary Supplement: A1PF milk consumption, and then conventional cow's milk consumption

INTERVENTIONS:
Other: Dietary Supplement: conventional cow's milk consumption, and then A1PF milk consumption — Milk was consumed three times per day after meals, with 250 mL provided at each administration. During washout periods, participants were required to avoid all dairy products and use only rice milk.
  Arms: Sequence 1
Other: Dietary Supplement: A1PF milk consumption, and then conventional cow's milk consumption — Milk was consumed three times per day after meals, with 250 mL provided at each administration. During washout periods, participants were required to avoid all dairy products and use only rice milk.
  Arms: Sequence 2

SUMMARY:
This was a single-site, double-blind, randomised, controlled, crossover study, which aimed to compare the effects of conventional cow's milk (CON, containing both A1- and A2-types of beta-casein) versus milk free of A1-type beta-casein (A1PF milk) on gastrointestinal (GI) physiology and symptoms of digestive discomfort in non-regular milk drinkers with self-reported intolerance to conventional cow's milk. The study location was the Pennington Biomedical Research Center in Louisiana, USA. The study comprised a 2-week washout period, 2 weeks of milk consumption, crossover, a second 2-week washout period, and a second 2-week period of milk consumption. Eligible participants were stratified by sex to achieve an approximate 1:1 male to female ratio and were randomised to receive conventional cow's milk (sequence 1) or A1PF milk (sequence 2) during the first period of milk consumption. During the second period of milk consumption, participant groups underwent crossover to receive the alternate study milk.

Milk was consumed three times per day after meals, with 250 mL provided at each administration. During washout periods, participants were required to avoid all dairy products and use only rice milk to replace any normal dairy intake, and to avoid foods with very high fermentable oligosaccharides, disaccharides, monosaccharides, and polyols content, to avoid potential confounding of the symptoms experienced. Any medication, nutritional supplements, dairy products, acidophilus milk, or probiotics were prohibited during the study.

The study protocol and all related documentation were approved by the Pennington Biomedical Research Center Institution Review Board. The study was conducted in accordance with the principles of the Declaration of Helsinki and the Good Clinical Practice Guidelines of the International Conference on Harmonisation. All participants provided written informed consent prior to initiating any study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 18 to 68 years
* Irregularly consumed milk
* Had self-reported mild-to-moderate digestive discomfort after milk consumption
* Had normal electrocardiograms and blood pressure during quiet respiration

Exclusion Criteria:

* Known allergies to dairy products
* Severe milk intolerance
* A history of faecal impaction
* Having suffered from GI disorders (e.g., irritable bowel syndrome, colitis, ulcerative colitis, or coeliac disease)
* Currently being administered drugs for cardiovascular or metabolic disease
* Trying to lose weight by following a diet or exercise regimen
* Took any appetite or weight loss drugs for the previous three months

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 54 (Actual)
Dates: Start 2017-04-28 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-03-27 (Actual)

PRIMARY OUTCOMES:
Severity of bloating, abdominal pain, gas, borborygmus, eructation, and diarrhoea measured via Visual Analogue Scale (VAS) | At day 28 and day 56 (day 1 is study start)
  VAS: 0 = never; 1 = rarely; 2 = frequently; 3 = all the time

OTHER OUTCOMES:
Gastric transit time, hours | At day 28 and day 56 (day 1 is study start)
Frequency of adverse events | From day 1 to day 56 (day 1 is study start)
  Record if an adverse event is singe or intermettent.
Blood immunoglobulin (Ig)G, mg/dL | At day 28 and day 56 (day 1 is study start)
Fecal beneficial short-chain fatty acids (SCFA), mmol/g | At day 28 and day 56 (day 1 is study start)
Intensity of adverse events | From day 1 to day 56 (day 1 is study start)
  Record if an adverse event is mild, moderate, or severe.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States